CLINICAL TRIAL: NCT06568419
Title: eBehandling - Health and Work Utility, Use and User Experience of a New Digital Transdiagnostic Work-Focused Intervention for Patients in Specialist Mental Health Care
Brief Title: eBehandling - Health and Work for Patients in Specialist Mental Health Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solli Distriktspsykiatriske Senter (Other)
Collaborators: Sykehuset Innlandet HF (Other); Sykehuset Ostfold (Other); Sykehuset i Vestfold HF (Other); University Hospital, Aker (Other); Helse Fonna (Other); Helse Bergen Hospital Trust (Unknown); Vestre Viken Hospital Trust (Other); Macquarie University, Australia (Other); Diakonhjemmet Hospital (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 733956
Record Dates: First submitted 2024-07-08; First posted 2024-08-23 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Depression
Keywords: Sick Leave; Absemteeism; Transdiagnostic treatment; Internet-based Cognitive Behavioural Therapy
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: a non-randomized, single arm, multi-center mixed methods clinical trial in a naturalistic setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital transdiagnostic work-focused CBT treatment program (Experimental): digital transdiagnostic work-focused CBT treatment program for patients with common mental health disorders on sick leave or work assessment allowance
  Interventions: Behavioral: Transdiagnostic, work-focused Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Transdiagnostic, work-focused Cognitive Behavioural Therapy — Transdiagnostic, work-focused Cognitive Behavioural Therapy focuses on core mechanisms that creates and maintain illness in depression and anxiety. Namely reducing avoidance and/or suppression of unwanted thoughts, avoidance of meaningful activity and increase cognitive flexibility while under psychological stress.

SUMMARY:
Mental health problems and disorders affect one in every five amongst the working- age adults in the countries of the Organization for Economic Cooperation and Development. This constitutes a major public health challenge that also has large implications for work participation and productivity.

Major depression and anxiety are the most prevalent of the mental disorders and are therefore named common mental disorders (CMD). CMD have become a major cause of work absenteeism, with 30% of all sick leave in Norway being due to CMDs in 2024.

Early interventions addressing psychological aspects and vocational challenges related to work have shown a positive effect on return to work. Therefore, finding ways to increase availability and reduce barriers to evidence-based treatments seems a viable route to reducing mental health's impact on sick leave and absenteeism.

Research show that improvement in symptoms from ordinary psychotherapy has little impact on sick-leave. The same results have been found for internet-based cognitive therapy (ICBT). One of the challenges in specialised mental health care is that the work focus has been an additive or extended part of the treatment, not integrated in the treatment itself.

Several studies have been conducted on psychological treatments that specifically target return to work for people with CMDs. Systematic reviews have shown that work-focused therapy has a small, but significant effect over treatment as usual on return to work and finds that 20% more workers in the intervention groups had returned to work, compared to control groups.

The availability of traditional therapy is scarce and there is an need for new effective ways of delivery. internet-based cognitive therapy has been shown to be as effective as traditional therapy in many systematic reviews and meta analysis and seems a good approach to reach the goal of increasing availability.

To account for the heterogene group of people on sick leave the investigators have created a transdiagnostic, work-focused internet-based cognitive behaviloural therapy program.

This study aims is to is to investigate the utility and use of this treatment program for patients with common mental health disorders on sick leave or work assessment allowance. This includes the user experience of participation and experienced utility of the treatment program.

DETAILED DESCRIPTION:
Study aims The main aim of the current study is to investigate the utility and use of a digital transdiagnostic work-focused CBT treatment program for patients with common mental health disorders on sick leave or work assessment allowance. This includes the user experience of participation and experienced utility of the treatment program. Secondary aims are related to mediators and moderators of treatment efficacy and the participants' experience with the program.

Research questions

1. To what extent does the treatment program impact Return to Work, self-reported symptoms, and everyday functioning?
2. To what extent do clinical, work-related and demographic factors affect treatment adherence and treatment response?
3. To what extent do adherence and changes in work-related self-efficacy predict outcomes?
4. What type and frequency of negative effects does participants report?
5. How do participants describe their experience of use and utility of the program, as well as its challenges and benefits?

   Hypotheses of main effects H1a. The investigators expect a large main effect of treatment on total percentage sick leave from pre- to post treatment, with gains maintained at follow up.

   H1b. The investigators expect a large main effect of treatment on the number of participants with full return to work from pre- to post treatment, with gains maintained at follow up.

   H2. The investigators expect a large main effect of treatment on reduction on symptoms of depression and anxiety.

   H3. The investigators expect a positive main effect of treatment on Return to Work Self-Efficacy, from pre to post treatment, and sustained through follow up.

   Hypotheses of moderating and mediating effects and predictors of outcome H4. The investigators expect a negative relationship between duration of baseline work absenteeism and degree of return to work at post. Baseline work absenteeism will moderate the relationship between treatment and return to work.

   H5a. The investigators expect treatment credibility at baseline to be predictive of treatment adherence.

   H5b. The investigators expect that treatment adherence will be a mediator between treatment credibility and treatment outcome.

   H6. The investigators expect changes on the Return to Work Self-Efficacy Scale to predict the degree of absenteeism post treatment.

   H7. The investigators expect change on the Return to Work Self-Efficacy Scale to be a mediator between baseline absenteeism and return to work post-treatment.

   H8. The investigators expect higher depression scores (PHQ-9/CORE-OM score) to be a moderator between treatment credibility and treatment outcome and adherence.

   H9. The investigators expect that fewer than 10% of participants experience negative effects caused by participation, as measured by the Negative Effects Questionnaire (NEQ).

   Measures

   Demographic variables. Self-reported data will be collected on gender, age, level of education, length and degree of sick leave, length of mental health problems and marital status.

   Primary and secondary F-diagnosis (ICD-10) will be reported by the eTherapist. Questionnaires.

   Primary outcome measures: The reduction in the degree of sick leave is one of our primary outcomes and will be measured through self-report.

   The Return to Work Self-Efficacy Scale

   Secondary outcome measures:

   The Generalized Anxiety Disorder-7

   The Patient Health Questionnaire-9

   The Work and Social Adjustment Scale

   CORE-OM

   CORE-10 The Negative Effects Questionnaire

   An adapted version of the Credibility Rating Scale

   System data on user behaviour. Data on use and user behaviour will be extracted from the system and combined with data from the self-report questionnaires collected. Information about the actual program use will be generated by the e-health platform Youwell. The data includes the extent to which participants complete the treatment, where and when the participants drop out, and how long the participants need to complete individual parts.

   Further The investigators also will analyse how long each session lasts and what system and platform the participants use. Each eBehandling location will also maintain local statistics on the number of assessment interviews, participants included and excluded to assess acceptance in the patient population and hospital setting.

   Qualitative in-depth interviews. Two months after completion of the program, a subset of participants will be invited to an in-depth interview. The investigators will use purposive sampling to select participants who represent a diverse range of demographics (age, gender) and outcomes (treatment responders and non-responders). The investigators aim to recruit a total of 20 participants for the qualitative interviews, likely ensuring richly-textured information on a broad array of participant experiences.

   The treatment intervention is a digital transdiagnostic work-focused cognitive behaviour therapy program. The program consists of seven modules consisting of psychoeducational texts, imagery and models, in addition to therapist-tailored tasks for the participants. The treatment model is based on traditional CBT principles and adjusted to target transdiagnostic maintaining mechanisms in anxiety and depression such as frequent negative emotions and aversive reactions to these that leads to various forms of avoidant coping that serve to reinforce the negative emotional cycle.

   Treatment will be given by trained eTherapists with specific training in the eBehandling - health and work protocol. Further the participants will be given a one-day introduction on the use of W-CBT within a digital format by the authors of the program.

   Quantitative analyses. In order to identify factors associated with treatment success and outcomes, hierarchical linear mixed modelling analyses (HLM, "multilevel") will be conducted. The models will be checked if the participants fulfil the model assumptions of normality of residuals, linearity and homoscedasticity. The dependent variables are sick leave, work related self-efficacy (as measured by RTWSE-11), depression severity (PHQ-9), anxiety (GAD-7), well-being, symptoms, risk and function (CORE-OM) and impairment in functioning (WSAS). The predictors are: Treatment (time), duration of sick-leave prior to treatment, treatment credibility, work related self-efficacy, depression severity and adherence. Comparisons are modelled through main effect and interaction effect analysis (e.g. Time x "Baseline work absenteeism" interaction). Predictors will be centred using grand mean centering. T-values and degrees of freedom will be estimated using "Sattertwaite" correction. The effects sizes will be converted from t-values and degrees of freedom to Cohen's d. Corrections for multiple analyses will be done by using Jaccard's correction to decrease risk of Type I error when applying several statistical tests.

   Qualitative analyses. Transcribed interviews will be analysed with the software NVivo 14 using reflexive thematic analysis. By comparing the individual accounts, The investigators want to identify both patterns of commonalities and differences in participants' experiences and formulate these as themes.

   Power analyses As stated by Van Voorhis and Morgan (2007): "if the circumstances allow, a researcher would have better power to detect a small effect size with approximately 30 participants per variable. Following this rule of thumb, The investigators plan for 30 participants per predictor (unique main effects), thus a total sample size of 300 participants. Calculating a drop-out rate of 30% gives a total sample size of N = 390.

   Procedure Inclusion will be open for 18 months, planned from September 2024. Participants will be recruited from outpatient specialised mental health care facilities in the Western Norway Regional Health Authority and South-Eastern Norway Regional Health Authority. After recruitment, each participant will undergo an assessment for eligibility where inclusion and exclusion criteria are evaluated. If eligible, participants are asked to sign a written informed consent to participation before enrolment in the study. Participants can at any time during treatment withdraw their consent. In this case the participants will be able to continue treatment, but their user data will not be exported for research purposes.

   The main form of contact between participant and eTherapist will be via asynchronous messages. If asked for by the participant, or evaluated as necessary by the eTherapist there will be contact via phone or face-to-face.

   After 12 weeks the participants will be given a concluding session face-to-face where the next step is decided: End treatment, further treatment within the specialist mental health care services or referred to a different treatment option. Regardless of this the participants will have access to the treatment program, without therapist contact, for six months after completion.

   Ethical considerations

   The therapist's level of competence

   The therapists giving the treatment program are clinical psychologists or have at least a bachelor degree in health. All therapists are trained in eTreatment in general, this program specifically and are given weekly or bi-weekly guidance on eTherapy within their workplace and by the project group.

   Monitoring suicidal risk or behaviour Participants will each week answer question 10 (suicidal ideations) of the Montgomery and Åsberg Depression Rating Scale and the total CORE-10. Both of these questionnaires have a cut-off for risk which, if surpassed, leads to an automatic text message and e-mail to the participants' eTherapist and local program supervisor. The eTherapist, or the program supervisor contacts the participant and follows their local procedure on assessing suicidal risk and take precautionary measures as deemed necessary.

   Transdiagnostic treatment for specific or comorbid diagnosis There is compelling evidence that transdiagnostic treatment protocols are effective in influencing the underlying mechanisms of CMDs through the reduction of fear and avoidance of-, and increasing acceptance of emotions, physical sensations and establishing alternative, more adaptive behaviours. This is found in both face-to-face therapy and ICBT. As The investigators have developed the treatment in the current study on these established principles The investigators see no imminent increased risk of reduced effect of the treatment on CMDs in this study.

   In the case of participant drop out If a patient drops out of treatment, or together with their eTherapist concludes that the treatment program of this study is not suitable, the participants will be given access to other, suitable treatment either via "eBehandling" or face-to-face treatment at their local District Psychiatric Center.

   Data and privacy protection The Youwell platform and concerns of health information have been processed and approved for clinical use via the Western Norway Regional Health Authority based on a risk and vulnerability analysis and Data Protection Impact Assessment

   Financing sources The study is currently funded by Solli DPS and previously assigned strategic funding from the Western Norwegian Regional Health Authority. The investigators will apply for funding from the Western Norwegian Regional Health Authority.

   Conflicts of interest No conflicts of interest are stated by the research project group.

ELIGIBILITY:
Inclusion Criteria:

1. being an outpatient in specialised mental health care service,
2. above 18 years old,
3. full or graded sick leave, or on work assessment allowance
4. primary diagnosis of F30 - F40 (ICD-10),
5. currently employed.

Exclusion Criteria:

1. ongoing psychotic disorder and/or mania,
2. ongoing substance abuse, incl. sedative medications,
3. ongoing episode of major depression,
4. organic brain disease,
5. severe reading and writing difficulties.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Degree of Sickleave | baseline, 6 weeks, 12 weeks, 6 months and 12 months
  Self-reported degree of sick leave (percentage)
Return to Work Self-efficacy 11 | baseline, 6 weeks, 12 weeks, 6 months and 12 months
  11-item questionnaire measuring an individual's confidence in their ability to work and perform work tasks. Items are scored on a scale from 1 ("Totally disagree") to 6 ("Totally agree"). Items 2 and 6 are reversed.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | baseline, 6 weeks, 12 weeks, 6 months and 12 months
  measure of worry and anxiety and consists of seven items scored from 0 ("Not at all") to 3 ("Nearly every day") and one additional item measuring how the symptoms affect functioning.
Patient Health Questionnaire-9 | baseline, 6 weeks, 12 weeks, 6 months and 12 months
  measures depression severity. The measure consists of nine items scored from 0 ("Not at all") to 3 ("Nearly every day").
The Work and Social Adjustment Scale | baseline, 6 weeks, 12 weeks, 6 months and 12 months
  measures impairment in functioning. The measure consists of five items scored from 0 (not at all impaired) to 8 (very severely impaired)
CORE-OM | baseline, 6 weeks, 12 weeks, 6 months and 12 months
  a 34-item self-report, measuring well-being, symptoms, elements of risk, and function on a five-point scale ranging from "not at all" to "most, or all the time".
CORE-10 | at 2, 4, 8 and 10 weeks
  a ten item self-report measuring symptoms, well-being, functioning and risk on a five-point scale ranging from "not at all" to "most, or all the time"
The Negative Effects Questionnaire | at 12 weeks
  a 20-item questionnaire evaluating adverse or unwanted events during treatment. Participants report whether a specific event occurred during treatment ("Yes"/"No") and then indicate how negatively they were affected by it on a scale ranging from 0-4.

OTHER OUTCOMES:
Credibility Rating Scale | baseline, 6 weeks and 12 weeks
  An adapted version of the Credibility Rating Scale (Borkovec & Nau 1972) will be used to assess treatment credibility. The scale consists of five items where participants rate their credibility/expectancy-for-improvement on a 10-point scale.
Montgomery and Åsberg Depression Rating Scale | baseline and every week for 12 weeks (until the end of the treatment program)
  Participants will each week answer question 10 (suicidal ideations)

CONTACTS AND LOCATIONS:
Overall Officials: Pål William Wallace, PhD, Study Director — Solli DPS; Kristine Sirevåg, MSc, Study Chair — Solli DPS
Locations (9):
- Norway (9):
  - Sykehuset Vestre Viken, Oslo, Bærum
  - Sykehuset Innlandet, Lillehammer, Innlandet
  - Sykehuset i Vestfold, Tønsberg, Vestfold
  - University of Bergen, Bergen, Vestland
  - Bjørgvin DPS (Helse Bergen), Bergen, Vestland
  - Solli DPS, Bergen, Vestland
  - Vinderen DPS, Oslo
  - AHus DPS Grorudalen, Oslo
  - Sykehuset i Østfold, Fredrikstad, Østfold fylke

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-06-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT06568419/Prot_000.pdf